CLINICAL TRIAL: NCT06161350
Title: The Multi-disciplinary Approach of Children With Feeding Difficulties and Tube Feeding in UZB Between 2000 and 2021: a Retrospective Cohort Study
Brief Title: The Multi-disciplinary Approach of Children With Feeding Difficulties and Tube Feeding in UZB Between 2000 and 2021
Acronym: ORALAV
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Elisabeth De Greef, Prof. Dr. De Greef, Universitair Ziekenhuis Brussel
Other Study IDs: ORALAV
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Oral Aversion; Enteral Nutrition; Parenteral Nutrition; Tube Feeding
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Infants who consulted between January 1st 2000 and December 31st 2009 (this is before the implementation of the pre-convention).
  Inclusion criteria:
  * Children consulting a pediatric gastroenterologist for feeding problems in UZB between the 1st of January 2000 and the 31st of December 2009 and receiving the label "feeding difficulties".
  * The infants have a pediatric feeding disorder that prevent them from feeding normally by oral means.
  * The infants need or have needed (enteral or parenteral) artificial nutrition.
  * The infants are aged between 0 and 12 years at their first presentation.
  * The infants are capable of developing normal feeding behavior.
  Infants will be excluded from this study if they:
  * Have no 6-months follow-up available.
  * Parents refusal to enter a multi-disciplinary approach for the feeding problems of their children.
- Group 2: Infants who consulted after the implementation of the pre-convention, who consulted between January 1st 2010 and December 31st 2021.
  Inclusion criteria:
  * Children consulting a pediatric gastroenterologist for feeding problems in UZB between the 1st of January 2010 and the 31st of December 2021 and receiving the label "feeding difficulties".
  * The infants have a pediatric feeding disorder that prevent them from feeding normally by oral means.
  * The infants need or have needed (enteral or parenteral) artificial nutrition.
  * The infants are aged between 0 and 12 years at their first presentation.
  * The infants are capable of developing normal feeding behavior.
  Infants will be excluded from this study if they:
  * Have no 6-months follow-up available.
  * Parents refusal to enter a multi-disciplinary approach for the feeding problems of their children.
  Interventions: Combination Product: Structured multi-disciplinary approach

INTERVENTIONS:
Combination Product: Structured multi-disciplinary approach — Since 2010, a structured multidisciplinary team was formed to evaluate the child medically, support its nutrition, teach, treat and educate the children and parents and guide them through the process to obtain a normal and independent feeding behavior. The multidisciplinary team must have special expertise regarding digestive and nutritional as well as sensory and oral motor problems in children requiring artificial nutrition. The team must at least consist of a pediatrician, a dietician with experience in artificial nutrition in children, a speech therapist and/or physical therapist and a psychologist or orthopedagogue. The team should also be able to rely on a nurse with experience in artificial nutrition, a social assistant and a secretary.
  Groups: Group 2

SUMMARY:
The goal of this Retrospective Cohort Study is to compare the patients from before and after the implementation of the pre-convention for infants with feeding difficulties needing tube feeding or having received tube feeding in the past, but able to develop normal feeding behavior.

The main objectives it aims to compare are:

* To characterize the patients taking part in a multi-disciplinary follow-up for feeding difficulties over time and to evaluate their progress before and after the institution of a multidisciplinary team in the context of the pre-convention for feeding difficulties from the RIZIV/INAMI.
* To evaluate if the multi-disciplinary approach is more efficient for treatment and follow-up in infants with eating difficulties before and after the start of the pre-convention.
* To calculate the probability of reaching full oral intake after having feeding difficulties within two years.

ELIGIBILITY:
Inclusion Criteria:

* Children consulting a pediatric gastroenterologist for feeding problems in UZB between the 1st of January 2000 and the 31st of December 2021 and receiving the label "feeding difficulties".

The infants have a pediatric feeding disorder that prevent them from feeding normally by oral means.

* The infants need or have needed (enteral or parenteral) artificial nutrition.
* The infants are aged between 0 and 12 years at their first presentation.
* The infants are capable of developing normal feeding behavior.

Exclusion Criteria:

* Have no 6-months follow-up available.
* Parents refusal to enter a multi-disciplinary approach for the feeding problems of their children.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with feeding difficulties needing tube feeding or having received tube feeding in the past, capable of developing normal feeding behavior.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Growth (weight-for-height Z-scores) | at 3, 6, 12, 18 months and 2 years

SECONDARY OUTCOMES:
Comparing the mean of the 2 groups of total number of days tube fed | At 3, 6, 12, 18 months and 2 years
Comparing the mean of the 2 groups of the percentage of intake through tube feeding | At 3, 6, 12, 18 months and 2 years

OTHER OUTCOMES:
Compare how many infants completed full oral intake after two years before and after the implementation of the pre-convention for feeding difficulties. | 2 years
Compare the percentage of tube feeding that remains in the group that was unable to achieve full oral intake after one year, before and after the implementation of the pre-convention for feeding difficulties. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth De Greef, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel; Koen Huysentruyt, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided